CLINICAL TRIAL: NCT07012837
Title: Reducing Point-of-Care Transfusion Requirements With Prolonged Desmopressin in High-Bleeding-Risk Cardiac Surgery: A Multicentre Randomized Controlled Trial (REDES-BLEED)
Brief Title: Transfusion Reduction in High-Bleeding-Risk Cardiac Surgery With Desmopressin
Acronym: REDES-BLEED
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Imam Abdulrahman Bin Faisal University (Other)
Collaborators: Johns Hopkins Aramco Healthcare (Other)
Responsible Party: Principal Investigator, Mohamed R El Tahan, Consultant in Cardiac Anesthesia, Imam Abdulrahman Bin Faisal University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: IABF-10-05-25
Record Dates: First submitted 2025-06-01; First posted 2025-06-10 (Actual); Last update posted 2025-06-10 (Actual); Status verified 2025-06

CONDITIONS: Adult Patients Undergoing Cardiac Surgery; High Bleeding Risks; Planned Elective Cardiac Surgery Using CPB
Keywords: Adult cardiac surgery; Cardiopulmonary bypass; High bleeding risks; Desmopressin; Prophylactic; Point-of-care coagulation tests

STUDY DESIGN:
Intervention Model Description: A multicenter, parallel, two-group, prospective, multicenter, randomized, blinded comparative trial in patients with high risks of postoperative bleeding scheduled for elective cardiac surgery at the King Fahad Hospital of Imam Abdulrahman Bin Faisal University, Al Khobar and Johns Hopkins Aramco Healthcare, Dhahran, Saudi Arabia.
Who Masked: Participant, Outcomes Assessor
Masking Description: Further minimization of bias will be achieved by involving two independent investigators. The researcher who is not responsible for providing anesthesia or performing surgery will perform the Randomization directly before the start of anesthesia. A second investigator, blinded for the randomization arm, will record the primary and secondary postoperative outcome measures.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Before induction of anesthesia, patients will receive identical and similar clear study solutions in similar size transparent 50-cc bags, including Saline will be infused over five hours at a rate of 10 ml/hr.
  The local pharmacists who will not be involved in patients' care or data collection will prepare the study solution.
  Interventions: Drug: Placebo
- Desmopressin (Active Comparator): Before induction of anesthesia, patients will receive identical and similar clear study solutions in similar size transparent 50-cc bags, including Desmopressin 0.3 ug/kg of the patient's body weight will be infused over five hours at a rate of 10 ml/hr. The local pharmacists who will not be involved in patients' care or data collection will prepare the study solution.
  Interventions: Drug: Desmopresin

INTERVENTIONS:
Drug: Placebo — Before induction of anesthesia, patients will receive identical and similar clear study solutions in similar size transparent 50-cc bags, including Saline will be infused over five hours at a rate of 10 ml/hr. The local pharmacists who will not be involved in patients' care or data collection will prepare the study solution.
  Arms: Placebo
Drug: Desmopresin — Before induction of anesthesia, patients will receive identical and similar clear study solutions in similar size transparent 50-cc bags, including Desmopressin 0.3 ug/kg of the patient's body weight will be infused over five hours at a rate of 10 ml/hr. The local pharmacists who will not be involved in patients' care or data collection will prepare the study solution.
  Arms: Desmopressin

SUMMARY:
Rationale

Bleeding after cardiac surgery is a complication that might result in increased morbidity, mortality, and cost of cardiac surgery by 1.76 (confidence interval (CI), 1.64-1.90) times and a median increase in costs by Australian $33,338 (CI, $21,943-$38,415) [1]. Strategies and techniques to reduce postoperative bleeding in identified high-risk patients for bleeding after cardiac surgery might improve outcomes and resource utilization.

Desmopressin (DDAVP) is used as a hemostatic agent to prevent and treat bleeding in patients with mild hemophilia patients with von Willebrand's deﬁciency through stimulating the release of von Willebrand factor from endothelial cells.

Previous studies showed controversial results in terms of reduced transfusion requirements in patients with low risk for bleeding with post cardiopulmonary bypass (CPB) bleeding following prophylactic infusing desmopressin over 10 to 15 minutes after induction of anesthesia or protamine administration due to its positive effects on the coagulation system responsible for such bleeding. Contradictory, prophylactic desmopressin use demonstrated fewer transfusion requirements in patients treated with antiplatelets, which raises the need to examine its efficacy in high-risk cardiac surgery patients for perioperative bleeding. These controversial results might be attributed to delayed administration of desmopressin after evolving CPB-associated thrombocytopenia, platelet dysfunction, coagulation factor consumption and dilution, hyperfibrinolysis, and hypofibrinogenemia [2]

Concerns were raised about the associated transient decreases in systemic vascular resistance and blood pressure after desmopressin administration following discontinuing CPB and administering protamine, which might be related to the rapid infusion rate during the critical surgery stage.

The cost of a single dose of Desmopressin 0.3 ug/kg for a patient with an average weight of 70 Kg is about 82US$ which is cheaper than the alternative hemostatic agents proved to be effective in reducing bleeding and transfusion needs after cardiac surgery (e.g., fibrinogen concrete (average of 3 g = 1,167US$) and prothrombin complex concentrate (6,255US$ considering low fixed dosfixed-doseof 1040 IU F IX).

It is yet unclear if extended infusions of desmopressin started earlier before the development of CPB-associated coagulopathy and platelets dysfunction from anesthesia induction time and continued to the end of CPB before protamine administration would offer an "efficacy," "safety, and "cost-effective" benefits over placebo in patients with high risks for bleeding after cardiac surgery terms of the need for transfusion, cumulative postoperative 48-hour chest tube outputs, need for reoperation, thrombotic complications, 30-day mortality, hemodynamic stability, and urine output during and after completing infusion, and costs of the study drug and allogenic transfusion requirement. That raises the need to examine its impact on these crucial clinical outcomes.

Objective

The primary objective of this prospective multicentre randomized clinical trial (RCT) is, compared with placebo, to examine the impact of prolonged infusion desmopressin on reducing postoperative bleeding and the need for allogenic allogeneic transfusion in high-bleeding-risk cardiac surgery patients scheduled for elective cardiac surgical procedures using CPB. Secondary objectives include comparing placebo and desmopressin in terms of safety and cost-effectiveness.

Hypothesis

It is hypothesized that extended 'desmopressin' infusion compared to 'placebo' results in less postoperative bleeding and transfusion needs (more effective) and leads to less hemodynamic compromise (safer) and cheaper (cost-effective) in high-risk cardiac surgery patients.

DETAILED DESCRIPTION:
3. INTRODUCTION AND RATIONALE

3.1 The current role of prophylactic use of desmopressin in low-risk cardiac surgery patients.

The efficacy of "routine prophylactic administration" of desmopressin 0.3 ug/kg after anesthesia induction or protamine administration to reduce bleeding and transfusion has been revisited in a Cochrane review of 39 randomized controlled trials (RCTs) focusing on cardiac surgery [5] which demonstrated that compared with placebo, desmopressin used resulted in a slight decreased total volume of red blood cells (RBCs) transfused (mean difference (MD) -0.52 units, 95%CI -0.96 to -0.08 units; 14 trials, 957 participants) and total blood loss (MD -135.24 mL, 95% CI -210.80 mL to -59.68 mL; 22 trials, 1,358 participants) in adult cardiac surgery. These RCTs had low methodological quality.

Desmopressin may reduce postoperative bleeding in cardiac surgery patients who have received preoperative aspirin within 7 days of surgery, longer cardiopulmonary bypass (CPB) bypass than 140 minutes, and those with platelet dysfunction [6].

A recent European Association for Cardio-Thoracic Surgery (EACTS) and the European Association of Cardiothoracic Anaesthesiology and Intensive Care (EACTAIC) guidelines on patient blood management (PBM) in adult cardiac surgery, in collaboration with the European Board of Cardiovascular Perfusion (EBCP), [7] concluded a task force of professionals specializing in patient blood management recommend that the prophylactic use of desmopressin is not recommended to reduce bleeding complications in cardiac surgery patients (a class III of recommendation and level A of evidence). However, it suggests considering desmopressin for bleeding patients with platelet dysfunction to reduce bleeding complications. (a class IIa of recommendation and level C of evidence).

3.2 Efficacy of Desmopressin in Reducing Postoperative Bleeding and Allogenic Blood Transfusion Needs

Although desmopressin showed a slight decrease in transfusion requirement in patients with post-CPB bleeding due to its positive effects on the coagulation system responsible for such bleeding, there is a continued debate on the "efficacy" and "safety" of prophylactic use of desmopressin for cardiac surgery [8-9].

A previous small study demonstrated the efficacy of desmopressin in reducing homologous blood requirement in cardiac surgical patients treated with aspirin within 5 days before surgery [10].

3.3. Does the timing of the Desmopressin Administration Make A Difference?

The timing of the administration of desmopressin might explain such controversial results. Infusing desmopressin following protamine administration failed to show significant differences in transfusion requirements in small studies, including few patients [11-13]. Similar results were reported when desmopressin was administered after chest closure [14]. Delaying desmopressin administration until the termination of CPB or chest closure, with its impact on the coagulation system and platelet functions, might explain these reported low or no efficacy in reducing bleeding compared with placebo. Additionally, this is contradictory to the highly recommended routine use of antifibrinolytics (class 1, Level of evidence A) and using protamine to heparin ratio of less than one (class 1, Level of evidence B) by the current EACTS/EACTAIC/EBCP Guidelines on PBM [6], that was not considered in these studies [10-14].

3.4. Can Repeating Desmopressin Administration Increase the Efficacy?

Repeating the administration of desmopressin after CPB and then 12 hours after surgery did not result in a significant difference despite the blood loss being less than that of the placebo in the former in a small, unpowered study [15-16].

3.5. Safety of Desmopressin Administration

Rapid infusing desmopressin over ten or 15 minutes, particularly shortly after administering protamine with its unique vasodilatation and histamine release effect, might explain the notable reduced systemic vascular resistance (SVR) and blood pressure and increased pulmonary vascular resistance (PVR) in some studies [10-14, 16], which was unlikely due to the associated histamine release [17].

Desmopressin use did not result in significant changes in urine output [12] or increased myocardial infarction incidence [15]; these studies included few patients to examine these secondary outcomes.

3.6. Can Slower Desmopressin Administration Increase Its Safety

A slower infusion of desmopressin over 30 rather than 10 minutes was only associated with less increased PVR in this small cohort [18]. That raises the need to examine the "safety" of a more extended infusion of desmopressin.

3.7. Can Point-of-Care Coagulation Testing Improve Efficacy of Desmopressin Administration

Point-of-care (POC) thromboelastography (TEG) guided hemostasis and transfusion reduced RBCs, plasma, and platelet transfusion, operating room (OR) length of stay (LOS), intensive care unit (ICU) LOS, and bleeding rate (P = 0.002) were reduced with compared with controls in a metanalysis include 9 RCTs, two of them on cardiac surgery patients [19]. However, that was not translated into associated reduced mortality rates [19].

Interestingly, a single-Canadian-center, retrospective, observational propensity-matched study demonstrated increased desmopressin administration after the introduction of point-of-care (POC) rotational thromboelastometry (ROTEM) testing with and associated statistically higher platelets transfusion [20].

3.8. Feasibility

Extended infusion of desmopressin from induction of anesthesia to the end of CPB has never been compared in terms of "efficacy," "safety," and "cost-effectiveness" in high-risk cardiac surgery patients for bleeding. Cardiac surgery in patients with a high risk for bleeding is more complex to perform, and it might take longer durations to be accomplished, increasing the overall healthcare costs, which could be unacceptable for the stakeholders. Using desmopressin infusion over a more extended period might be an "effective," "safe," and "affordable" choice.

3.6. Why this randomized clinical trial?

Infusing the same desmopressin dose of 0.3 ug/kg over a more extended duration from anesthesia induction until before administering protamine might have its potential benefits and disadvantages in patients with higher risks for bleeding. The proposed randomized clinical trial here will compare extended intraoperative infusion of 'desmopressin' with 'placebo' procedures concerning effects on cumulative blood loss, need for allogenic blood transfusion, and hemostatic drugs and their overall costs, safety, and feasibility. If 'desmopressin' is more effective and less safe and is cost-effective than the "placebo,' it should be used in this group of patients. If 'desmopressin' is comparable and less safe than the "placebo,' it should not be used in this group of patients.

ELIGIBILITY:
Inclusion Criteria:

* Adult 18 years or older.
* Scheduled for any type of elective cardiac surgery.
* Using CPB.
* General anesthesia is provided in an endotracheally intubated patient.
* A high risk of postoperative bleeding is defined as any of the following [21-23];

  * Redo or repeated surgery.
  * Treatment with platelet P2Y12 receptor--inhibiting drugs was discontinued for 7 days (ticlopidine, clopidogrel, and prasugrel) or 5 days (ticagrelor).
  * Any known coagulation disorders.
  * Hypofibrinogenemia less than 150 mg/dl.
  * Platelet count <100.000 cells/μL.
  * Chronic renal failure, whether dialysis-dependent or not.
  * Liver cell failure Child-Pugh class B or C or the Model for End-Stage Liver Disease (MELD) >=29
  * Infective endocarditis.
  * Acute type-A aortic dissection.
  * Expected surgery with CPB time longer than 150 minutes.
  * Preoperative estimated Papworth Bleeding Risk Score of 8% or greater [23].

Exclusion Criteria:

* Planned for cardiac surgery without CPB;
* Planned for a combined coronary revascularization surgery and a valve or intra-cardiac surgery;
* Pregnancy;
* Consent for another interventional study during anesthesia;
* No written informed consent;
* Preoperative need for mechanical circulatory support;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Estimated)
Dates: Start 2025-07 (Estimated); Primary Completion 2027-07 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Cumulative 48-hour postoperative bleeding | Intraoperative and for 48 hours after surgery
  The primary outcome is the cumulative 48-hour postoperative bleeding, defined as the sum of estimated intraoperative salvaged blood and blood loss and postoperative chest tube output for 48 hours from surgery.
  Intraoperative blood loss was calculated from the total volume in suction bottles (minus the volume of irrigating solution), weighed sponges, and the volume collected in the Cell-Saver reservoir (minus the volume of anticoagulant solution).
  After the chest is closed, hourly postoperative blood loss will be calculated from the chest tubes and drain reservoirs.

SECONDARY OUTCOMES:
The need for allogenic PRBCs transfusion | For 7 days after surgery
  the need for allogenic PRBCs transfusion during 7 days after surgery (and timings).
The need for allogenic transfusion of fresh frozen plasma | For the first 7 days after surgery
  The need for allogenic transfusion of fresh frozen plasma during the first 7 days after surgery (and timings).
The need for allogenic individual and pooled platelet units | For the first 7 days after surgery
  Allogenic individual and pooled platelet units needed to be transfused during the first 7 days after surgery (and timings).
The need for allogenic cryoprecipitates units | For the first 7 days after surgery
  Allogenic cryoprecipitates units needed to be transfused during the first 7 days after surgery (and timings).
The need for Recombinant Factor VIII administration | For the first 7 days after surgery
  Recombinant Factor VIII administration needed to be transfused during the first 7 days after surgery (and timings).
The need for fibrongoen concentrate (FC) administration | For the first 7 days after surgery
  F.C. administration needed to be transfused during the first 7 days after surgery (and timings).
The need for prothrombin complex concentrate (PCC) administration | For the first 7 days after surgery
  PCC administration needed to be transfused during the first 7 days after surgery (and timings).
Intraoperative urine output volume | Intraopertively
  Intraoperative urine output volume in ml.
The number of intraoperative hypotension episodes | Intraoperatively
  The number of intraoperative hypotension episodes unrelated to the surgical procedure step defined as a 15% decrease in mean arterial blood pressure (MAP) from baseline values lasted for 5 minutes and required intervention (e.g., fluid therapy, vasopressor, or inotropes as per the discretion of anesthesia provider).
Timings of intraoperative hypotension episodes | Intraoperatively
  Timings of intraoperative hypotension episodes in relation to study solution or protamine administration.
Intraoperative fluid balance | Intraoperatively
  Intraoperative fluid balance is the net of differences between intake and output during surgery.
The 24-hour fluid balance | For 24 hour after surgery
  The 24-hour fluid balance is defined as the net of differences between intake and output 24 hours after surgery.
The 48-hour fluid balance | For 48 hour after surgery
  The 48-hour fluid balance is defined as the net of differences between intake and output 48 hours after surgery.
The need for re-explorative surgery | For 30 days after surgery
  The need for re-explorative surgery during the same admission.
Postoperative ICU lenght of stay (LOS) | For 90 days after surgery
  Postoperative ICU LOS of days from the date of surgery until discharge from the ICU or death.
Postoperative hospital length of stay (LOS) | For 180 days after surgery
  Postoperative hospital LOS from the date of surgery until discharge from the hospital or death.
Postoperative documented death from a cardiovascular cause | For 30 days after surgery
  Postoperative documented death from a cardiovascular cause within 30 days of surgery.
Postoperative documented stroke | For 30 days after surgery
  Postoperative documented nonfatal stroke within 30 days of surgery.
Postoperative documented nonfatal myocardial infarction (MI) | For 30 days after surgery
  Postoperative documented nonfatal MI within 30 days of surgery.
Postoperative documented acute kidney injury (AKI) | For 7 days after surgery
  Postoperative documented AKI within 7 days of surgery.
Postoperative pulmonary complications | For 7 days after surgery
  Postoperative pulmonary complications are defined according to the PROVHILO study within 7 days of surgery
The overall costs of used desmopressin, allogenic blood units, and hemostatic drugs | For 180 days after surgery
  The overall costs of used desmopressin, allogenic blood units, and hemostatic drugs are represented in US$ as reported by the local pharmacy department.
Coronary graft thrombosis | For 3 months after surgery.
  Any documented coronary graft thrombosis within 3 months of surgery.
The need for revascularization | For 3 months after surgery.
  Any documented need for revascularization within 3 months of surgery.
Need for hospital re-admission at 30 days after surgery | For 30 days after surgery.
  Need for hospital re-admission at 30 days after surgery.
Need for hospital re-admission at 3 months after surgery | For 3 months after surgery.
  Need for hospital re-admission at 3 months after surgery.
Mortality at 30 days after surgery. | For 30 days after surgery
  Mortality at 30 days after surgery.
Mortality at 90 days after surgery. | For 90 days after surgery
  Mortality at 90 days after surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed R El Tahan, MD, Study Chair — Imam Abdulrahman Bin Faisal University; Fahad Makhdoum, MD, Principal Investigator — Imam Abdulrahman Bin Faisal University; Yasser F ElGhoneimy, MD, Study Director — Imam Abdulrahman Bin Faisal University
Locations (1):
- Imam Abdulrahamn Bin Faisal University (Former, Dammam University), Dammam, Eastern Province, Saudi Arabia

IPD SHARING:
Plan to Share IPD: Yes
The study database will be locked upon completion of data entry and resolution of all discrepancies or missing data, or when the investigators determine that no further resolution is feasible despite reasonable efforts. Prior to locking, a final review of the database will be conducted. Once locked, the dataset will be exported for statistical analysis.
  De-identified individual participant data (IPD), the study protocol, and statistical analysis plan will be made available upon reasonable request from qualified researchers beginning six months after publication and for a period of five years. Data access will be granted following review and approval of a research proposal and the signing of a data access agreement. Requests should be directed to the corresponding author.
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: Beginning six months after publication and for a period of five years.
Access Criteria: Data access will be granted following review and approval of a research proposal and the signing of a data access agreement. Requests should be directed to the corresponding author.

REFERENCES:
- [Background] Redfern RE, Fleming K, March RL, Bobulski N, Kuehne M, Chen JT, Moront M. Thrombelastography-Directed Transfusion in Cardiac Surgery: Impact on Postoperative Outcomes. Ann Thorac Surg. 2019 May;107(5):1313-1318. doi: 10.1016/j.athoracsur.2019.01.018. Epub 2019 Feb 12. PMID 30768933
- [Background] Khalil MA, El Tahan MR, Khidr AM, Fallatah S, Abohamar AD, Amer MM, Makhdom F, El Ghoneimy Y, Al Bassam B, Alghamdi T, Abdulfattah D. Effects of norepinephrine infusion during cardiopulmonary bypass on perioperative changes in lactic acid level (Norcal). Perfusion. 2023 Nov;38(8):1584-1599. doi: 10.1177/02676591221122350. Epub 2022 Aug 22. PMID 35994013
- [Background] Vuylsteke A, Pagel C, Gerrard C, Reddy B, Nashef S, Aldam P, Utley M. The Papworth Bleeding Risk Score: a stratification scheme for identifying cardiac surgery patients at risk of excessive early postoperative bleeding. Eur J Cardiothorac Surg. 2011 Jun;39(6):924-30. doi: 10.1016/j.ejcts.2010.10.003. Epub 2010 Nov 19. PMID 21094051
- [Background] Petricevic M, Petricevic M, Pasalic M, Golubic Cepulic B, Raos M, Vasicek V, Goerlinger K, Rotim K, Gasparovic H, Biocina B. Bleeding risk stratification in coronary artery surgery: the should-not-bleed score. J Cardiothorac Surg. 2021 Apr 21;16(1):103. doi: 10.1186/s13019-021-01473-3. PMID 33882969
- [Background] Baryshnikova E, Di Dedda U, Ranucci M. Are Viscoelastic Tests Clinically Useful to Identify Platelet-Dependent Bleeding in High-Risk Cardiac Surgery Patients? Anesth Analg. 2022 Dec 1;135(6):1198-1206. doi: 10.1213/ANE.0000000000006231. Epub 2022 Oct 13. PMID 36227767
- [Background] Orlov D, McCluskey SA, Callum J, Rao V, Moreno J, Karkouti K. Utilization and Effectiveness of Desmopressin Acetate After Cardiac Surgery Supplemented With Point-of-Care Hemostatic Testing: A Propensity-Score-Matched Analysis. J Cardiothorac Vasc Anesth. 2017 Jun;31(3):883-895. doi: 10.1053/j.jvca.2016.11.022. Epub 2016 Nov 17. PMID 28169116
- [Background] Dias JD, Sauaia A, Achneck HE, Hartmann J, Moore EE. Thromboelastography-guided therapy improves patient blood management and certain clinical outcomes in elective cardiac and liver surgery and emergency resuscitation: A systematic review and analysis. J Thromb Haemost. 2019 Jun;17(6):984-994. doi: 10.1111/jth.14447. Epub 2019 May 13. PMID 30947389
- [Background] Fleming NW, Burke TA. Infusion rate and hemodynamics with desmopressin. J Cardiothorac Anesth. 1989 Dec;3(6):813-5. doi: 10.1016/s0888-6296(89)96804-x. No abstract available. PMID 2521042
- [Background] Jahr JS, Marquez J, Cottington E, Cook DR. Hemodynamic performance and histamine levels after desmopressin acetate administration following cardiopulmonary bypass in adult patients. J Cardiothorac Vasc Anesth. 1991 Apr;5(2):139-41. doi: 10.1016/1053-0770(91)90326-o. PMID 1863724
- [Background] 16. Spyridakis, E., Pentilas, N., Retzios, G., Pappa, E., & Kalakonas, S. (2017). The use of desmopressin (DDAVP) as haemostatic agent in patients undergoing coronary artery bypass grafting (CABG) surgery. Journal of Cardiothoracic and Vascular Anesthesia, 31, S69.https://doi.org/10.1053/j.jvca.2017.02.153
- [Background] Marquez J, Koehler S, Strelec SR, Benckart DH, Spero JA, Cottington EM, Torpey DJ Jr. Repeated dose administration of desmopressin acetate in uncomplicated cardiac surgery: a prospective, blinded, randomized study. J Cardiothorac Vasc Anesth. 1992 Dec;6(6):674-6. doi: 10.1016/1053-0770(92)90049-d. PMID 1472662
- [Background] Salmenpera M, Kuitunen A, Hynynen M, Heinonen J. Hemodynamic responses to desmopressin acetate after CABG: a double-blind trial. J Cardiothorac Vasc Anesth. 1991 Apr;5(2):146-9. doi: 10.1016/1053-0770(91)90328-q. PMID 1863726
- [Background] Oliver WC Jr, Santrach PJ, Danielson GK, Nuttall GA, Schroeder DR, Ereth MH. Desmopressin does not reduce bleeding and transfusion requirements in congenital heart operations. Ann Thorac Surg. 2000 Dec;70(6):1923-30. doi: 10.1016/s0003-4975(00)02176-7. PMID 11156096
- [Background] Reich DL, Hammerschlag BC, Rand JH, Weiss-Bloom L, Perucho H, Galla J, Thys DM. Desmopressin acetate is a mild vasodilator that does not reduce blood loss in uncomplicated cardiac surgical procedures. J Cardiothorac Vasc Anesth. 1991 Apr;5(2):142-5. doi: 10.1016/1053-0770(91)90327-p. PMID 1863725
- [Background] Brown MR, Swygert TH, Whitten CW, Hebeler R. Desmopressin acetate following cardiopulmonary bypass: evaluation of coagulation parameters. J Cardiothorac Anesth. 1989 Dec;3(6):726-9. doi: 10.1016/s0888-6296(89)94790-x. PMID 2521029
- [Background] Dilthey G, Dietrich W, Spannagl M, Richter JA. Influence of desmopressin acetate on homologous blood requirements in cardiac surgical patients pretreated with aspirin. J Cardiothorac Vasc Anesth. 1993 Aug;7(4):425-30. doi: 10.1016/1053-0770(93)90164-g. PMID 8400098
- [Background] Hackmann T, Naiman SC. Con: desmopressin is not of value in the treatment of post-cardiopulmonary bypass bleeding. J Cardiothorac Vasc Anesth. 1991 Jun;5(3):290-3. doi: 10.1016/1053-0770(91)90291-z. PMID 1863751
- [Background] Shiffrin JS, Glass DD. Pro: desmopressin is of value in the treatment of post-cardiopulmonary bypass bleeding. J Cardiothorac Vasc Anesth. 1991 Jun;5(3):285-9. doi: 10.1016/1053-0770(91)90290-a. No abstract available. PMID 1863750
- [Background] 7. Casselman FPA, Lance MD, Ahmed A, Ascari A, Blanco-Morillo J, Bolliger D, Eid M, Erdoes G, Haumann RG, Jeppsson A, van der Merwe HJ, Ortmann E, Petricevic M, Weltert LP, Milojevic M; EACTS/EACTAIC/EBCP Scientific Document Group. 2024 EACTS/EACTAIC Guidelines on patient blood management in adult cardiac surgery in collaboration with EBCP. Interdiscip Cardiovasc Thorac Surg. 2024 Oct 10:ivae170. doi: 10.1093/icvts/ivae170. Epub ahead of print. PMID: 39385501.
- [Background] Wademan BH, Galvin SD. Desmopressin for reducing postoperative blood loss and transfusion requirements following cardiac surgery in adults. Interact Cardiovasc Thorac Surg. 2014 Mar;18(3):360-70. doi: 10.1093/icvts/ivt491. Epub 2013 Nov 21. PMID 24263581
- [Background] Desborough MJ, Oakland K, Brierley C, Bennett S, Doree C, Trivella M, Hopewell S, Stanworth SJ, Estcourt LJ. Desmopressin use for minimising perioperative blood transfusion. Cochrane Database Syst Rev. 2017 Jul 10;7(7):CD001884. doi: 10.1002/14651858.CD001884.pub3. PMID 28691229
- [Background] PROVE Network Investigators for the Clinical Trial Network of the European Society of Anaesthesiology; Hemmes SN, Gama de Abreu M, Pelosi P, Schultz MJ. High versus low positive end-expiratory pressure during general anaesthesia for open abdominal surgery (PROVHILO trial): a multicentre randomised controlled trial. Lancet. 2014 Aug 9;384(9942):495-503. doi: 10.1016/S0140-6736(14)60416-5. Epub 2014 Jun 2. PMID 24894577
- [Background] Smilowitz NR, Gupta N, Ramakrishna H, Guo Y, Berger JS, Bangalore S. Perioperative Major Adverse Cardiovascular and Cerebrovascular Events Associated With Noncardiac Surgery. JAMA Cardiol. 2017 Feb 1;2(2):181-187. doi: 10.1001/jamacardio.2016.4792. PMID 28030663
- [Background] Thiele RH, Raphael J. A 2014 Update on Coagulation Management for Cardiopulmonary Bypass. Semin Cardiothorac Vasc Anesth. 2014 Jun;18(2):177-89. doi: 10.1177/1089253214534782. PMID 24876232
- [Background] Newcomb AE, Dignan R, McElduff P, Pearse EJ, Bannon P. Bleeding After Cardiac Surgery Is Associated With an Increase in the Total Cost of the Hospital Stay. Ann Thorac Surg. 2020 Apr;109(4):1069-1078. doi: 10.1016/j.athoracsur.2019.11.019. Epub 2020 Jan 2. PMID 31904370